CLINICAL TRIAL: NCT07092969
Title: Comparison of the Effects of Aerobic and Anaerobic Exercises on Hormonal and Immune Biomarkers Measured by Blood and Saliva in Young Individuals
Brief Title: Comparison of the Effects of Aerobic-Anaerobic Exercises on Hormonal and Immune Biomarkers
Acronym: Biomarkers
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sakarya Applied Sciences University (Other)
Responsible Party: Principal Investigator, Abdurrahim Yıldız, Doç.Dr, Sakarya Applied Sciences University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2; 308-2025 (Other Grant/Funding Number: Sakarya BAP)
Record Dates: First submitted 2025-07-21; First posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Activity, Motor; Biomarkers; Exercise; Immunity
Keywords: Exercise physiology; Aerobic and anaerobic exercis; Hormonal and immunological responses; Physical activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: The study will be conducted in 2025 with 90 voluntary university students from the Department of Physiotherapy and Rehabilitation at Sakarya University of Applied Sciences. Participants will be aged 18-25 and free of chronic illnesses. Inclusion criteria are being a university student and within the specified age range. Exclusion criteria include orthopedic, cognitive, mental health problems, or chronic systemic diseases. Eligible students will be informed about the study's purpose, duration, potential risks, and methods, and will sign informed consent. Participants will be randomly divided into three equal groups, each receiving a different intervention, allowing comparison of physiological responses across groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group I - Control Group: (No Intervention): This group will not receive any training intervention. Participants will only undergo the Bruce Protocol and Wingate tests to serve as a baseline reference for physiological responses, allowing comparison with the other two groups.
- Group II - Treadmill Exercise (Bruce Protocol): (Experimental): Participants will perform the Bruce Protocol on a treadmill, which involves progressive stages of increasing speed and incline to challenge cardiovascular endurance. At each stage, heart rate, blood pressure, and fatigue level will be recorded. The session will end with a cool-down phase.
  Interventions: Device: Treadmill Exercise
- Group III - Bicycle Exercise (Wingate Anaerobic Test): (Experimental): This group will perform the Wingate Anaerobic Test using a stationary exercise bike. Following a warm-up, participants will cycle at maximum effort for 30 seconds to assess anaerobic performance. Data collected will include pedaling speed, power output, heart rate, and oxygen saturation.
  Interventions: Device: Bicycle Exercise

INTERVENTIONS:
Device: Treadmill Exercise — Participants in this group will perform an aerobic exercise using the Bruce Protocol on a treadmill. The test involves walking or running with gradually increasing speed and incline in predefined stages to assess cardiovascular endurance. Heart rate, blood pressure, and fatigue levels will be recorded at each stage. The session will conclude with a low-intensity cool-down phase.
  Arms: Group II - Treadmill Exercise (Bruce Protocol):
Device: Bicycle Exercise — The Wingate Anaerobic Test will be conducted using an ergometer bike. After a standardized warm-up, participants will pedal all-out for 30 seconds against a preset resistance, aiming to evaluate their anaerobic performance. Physiological parameters including power output, heart rate, and oxygen saturation will be monitored throughout the test.
  Arms: Group III - Bicycle Exercise (Wingate Anaerobic Test):

SUMMARY:
This study aims to compare the effects of aerobic and anaerobic exercise on hormonal, immunological, and metabolic biomarkers in young individuals using blood and saliva samples. It will also assess participants' physical activity levels, depression levels, and general lifestyle habits to explore their relationship with biomarker profiles. Biomarkers such as testosterone, progesterone, cortisol, IgA, alpha-amylase, insulin, lactate, and various inflammatory cytokines will be measured using ELISA. The study seeks to evaluate the physiological and psychosocial effects of different types of exercise in a holistic manner.

DETAILED DESCRIPTION:
Exercise is a complex stimulus that induces multifaceted effects on an individual's physiological and psychological systems. Aerobic and anaerobic types of exercise differ in terms of their energy production pathways and metabolic responses in the body. Aerobic exercises are long-duration, oxygen-dependent activities, while anaerobic exercises are short-duration, high-intensity activities that activate oxygen-independent energy systems.

These types of exercise cause various hormonal, immunological, and metabolic changes in the body. After exercise, significant changes are observed in biomarkers such as stress hormones (cortisol, progesterone), anabolic hormones (testosterone), immune system markers (IgA, TNF-α, IL-6, IL-10, IL-1β, IL-1RA, IL-4), and metabolic parameters (amylase, insulin, lactate). The fact that these parameters can be measured from both blood and saliva samples has increased the use of non-invasive methods in exercise physiology studies.

The level of physical activity is directly related not only to biological systems but also to an individual's psychological health and lifestyle habits. Research shows that regular physical activity reduces levels of depression and improves quality of life. The positive effects of exercise on the immune system become more significant when considered in conjunction with an individual's general lifestyle habits (nutrition, sleep, stress levels, substance use, etc.). It is particularly known that individuals with depression have high cortisol levels and suppressed IgA levels. Therefore, depression levels and lifestyle habits are important variables that affect the physiological responses to exercise.

This study will compare the effects of aerobic and anaerobic exercise on hormonal, immunological, and metabolic biomarkers measured via blood and saliva samples in young individuals. Additionally, the participants' physical activity levels, depression levels, and general lifestyle habits will be evaluated to explore the relationship between these variables and biomarker profiles. Measurements will include levels of testosterone, progesterone, cortisol, IgA, alpha-amylase, insulin, lactate, and various inflammatory cytokines, assessed using the ELISA method. In this way, the biological effects of different types of exercise will be evaluated from both physiological and psychosocial perspectives.

The main aim of this study is to comparatively examine the effects of aerobic and anaerobic exercises on hormonal, immunological, and metabolic biomarkers measured through blood and saliva samples in young individuals. Additionally, the relationship between the participants' physical activity level, depression level, and general lifestyle habits (nutrition, sleep patterns, substance use, etc.) with these biomarkers will be investigated, as well as the potential modulatory effects on the physiological responses to exercise.

ELIGIBILITY:
Inclusion Criteria:

* Being a university student,
* Being between the ages of 18 and 25.

Exclusion Criteria:

* Having orthopedic problems that prevent exercise,
* Having cognitive or mental health problems that prevent participation in exercise,
* Having chronic systemic diseases such as cardiac, pulmonary, or nephrological.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-09-15 (Estimated)

PRIMARY OUTCOMES:
Change in Salivary Testosterone Level | Time Frame: Baseline and immediately post-exercise Unit of Measure: pg/mL
  Measurement of testosterone concentration in saliva pre- and post-exercise.
Change in Salivary Cortisol Level | Time Frame: Baseline (pre-exercise) and immediately post-exercise (within 1 hour) Unit of Measure: ng/mL
  Measurement of cortisol concentration in saliva before and after aerobic and anaerobic exercise protocols.
Change in Salivary Progesterone Level | Time Frame: Baseline and immediately post-exercise Unit of Measure: pg/mL
  Salivary progesterone levels before and after exercise.
Change in Salivary Alpha-Amylase Activity | Time Frame: Baseline and post-exercise Unit of Measure: U/mL
  Enzymatic activity of salivary alpha-amylase as a stress marker.
Change in Blood Lactate Level | Time Frame: Baseline and post-exercise Unit of Measure: µIU/mL
  Lactate concentration in blood samples collected before and after exercise.
Change in Serum Cytokine Levels (e.g., IL-6, TNF-α) | Time Frame: Baseline and immediately post-exercise Unit of Measure: pg/mL
  Evaluation of pro- and anti-inflammatory cytokines in serum.
Change in Salivary Immunoglobulin A (IgA) | Time Frame: Baseline and post-exercise Unit of Measure: µg/mL
  Level of IgA in saliva as a marker of mucosal immune response.

SECONDARY OUTCOMES:
Change in Depression Score (Beck Depression Inventory-II) | Time Frame: Baseline (pre-intervention) and post-intervention (within 1 hour after final session) Unit of Measure: Score (range: 0-63) Method of Measurement: Self-reported questionnaire
  Assessment of participants' depressive symptoms using the validated Beck Depression Inventory-II (BDI-II).
Change in Physical Activity Level (IPAQ-Short Form) | Time Frame: Baseline and post-intervention Unit of Measure: MET-minutes/week
  Evaluation of participants' physical activity levels using the International Physical Activity Questionnaire - Short Form (IPAQ-SF), which estimates physical activity over the last 7 days in MET-minutes/week.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guest NS, VanDusseldorp TA, Nelson MT, Grgic J, Schoenfeld BJ, Jenkins NDM, Arent SM, Antonio J, Stout JR, Trexler ET, Smith-Ryan AE, Goldstein ER, Kalman DS, Campbell BI. International society of sports nutrition position stand: caffeine and exercise performance. J Int Soc Sports Nutr. 2021 Jan 2;18(1):1. doi: 10.1186/s12970-020-00383-4. PMID 33388079
- [Background] Pedersen BK, Hoffman-Goetz L. Exercise and the immune system: regulation, integration, and adaptation. Physiol Rev. 2000 Jul;80(3):1055-81. doi: 10.1152/physrev.2000.80.3.1055. PMID 10893431
- [Background] Gleeson M. Immune function in sport and exercise. J Appl Physiol (1985). 2007 Aug;103(2):693-9. doi: 10.1152/japplphysiol.00008.2007. Epub 2007 Feb 15. PMID 17303714
- [Background] Mikkelsen K, Stojanovska L, Polenakovic M, Bosevski M, Apostolopoulos V. Exercise and mental health. Maturitas. 2017 Dec;106:48-56. doi: 10.1016/j.maturitas.2017.09.003. Epub 2017 Sep 7. PMID 29150166
- [Background] Schuch FB, Vancampfort D, Firth J, Rosenbaum S, Ward PB, Silva ES, Hallgren M, Ponce De Leon A, Dunn AL, Deslandes AC, Fleck MP, Carvalho AF, Stubbs B. Physical Activity and Incident Depression: A Meta-Analysis of Prospective Cohort Studies. Am J Psychiatry. 2018 Jul 1;175(7):631-648. doi: 10.1176/appi.ajp.2018.17111194. Epub 2018 Apr 25. PMID 29690792